CLINICAL TRIAL: NCT05026268
Title: The Laparoscopic Right Colectomy With Intracoroporeal Anastomosis
Acronym: LaRCIa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/21
Record Dates: First submitted 2021-08-06; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Colon Cancer
Keywords: right colon cancer; laparoscopic right colectomy; intracorporeal anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomosis (Experimental): A laparoscopic right colectomy will be performed according to the surgeons standard practice with the intracorporeal anastomosis performing.
  Interventions: Procedure: intracorporeal anastomosis
- extracorporeal anastomosis (No Intervention): A laparoscopic right colectomy will be performed according to the surgeons standard practice.

INTERVENTIONS:
Procedure: intracorporeal anastomosis — intracorporeal stapled "side-to-side" isoperistaltic anastomosis
  Arms: Intracorporeal anastomosis

SUMMARY:
This is a randomized, controlled, "non-inferiority" trial to determine the non-difference in post-operative complications rate in laparoscopic right colectomy with intracorporeal or extracorporeal anastomosis formation.

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to laparosopic colectomy with intracorporeal or extracorporeal anastomosis.

Postoperative complications in both groups will be recorded in accordance with the Clavien-Dindo classification. The level of postoperative pain will be registred according to the visual analogue pain scale (VAS). Also the investigators will study the time of activation of patients, patient self-care scope according to the Bartell scale, postoperative hospital stay will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients age is 18 years and older
* Patients with right colon cancer
* Informed agreement

Exclusion Criteria:

* Carcinomatosis
* Primary tumor stage T4b
* Refusal of anastomosis
* Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications rate | 0 to 30 days
  The incidence and structure of postoperative complications according to the Clavien-Dindo scale (I-grade - any deviation from the normal course of the postoperative course without the need for pharmacological, surgical, endoscopic or interventional radiological interventions. drugs that are acceptable include antiemetics, antipyretics, analgesics, diuretics, and electrolytes. In addition, this grade includes a wound infection "stopped at the patient's bedside", V grades - Death of the patient).

SECONDARY OUTCOMES:
The level of postoperative pain | 0 to 10 days
  The level of postoperative pain with using a visual analogue pain scale: The patient assesses the postoperative pain from 0 to 10 points (0 points - no pain, 10 - unbearable pain).
The time of activation of patients | 0 to 10 days
  We will estimate time to verticalization of patients.
The amount of self-help of patients | 0 to 10 days
  We will estimate the amount of self-help of patients on the Bartel scale. Total score - 100. Indicators from 0 to 20 points correspond to complete dependence, from 21 to 60 points - severe dependence, from 61 to 90 points - moderate, from 91 to 99 life points - light dependence in everyday life.
The time to discharge from hospital | 0 to 30 days
  We will count days of postoperativa hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Russian Federation, Moscow, Russia